CLINICAL TRIAL: NCT01262599
Title: Effect of Pulsed Electromagnetic Fields on Postoperative Recovery After TRAM Flap Breast Reconstruction
Brief Title: Use of Pulsed Electromagnetic Fields (PEMF) After Breast Reconstruction Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Christine Hsu Rohde, MD, Assistant Professor of Clinical Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAE8848
Record Dates: First submitted 2010-12-01; First posted 2010-12-17 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Other Reconstructive Surgery
Keywords: Breast and abdomen morbidities after TRAM flap surgery; TRAM flap surgery; Post-mastectomy breast reconstructive surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham PEMF Device (Sham Comparator): Patients will receive inactive device
  Interventions: Device: Sham PEMF Device
- PEMF Device (Active Comparator): Patients will receive Ivivi Torino II PEMF Device
  Interventions: Device: Ivivi Torino II PEMF Device

INTERVENTIONS:
Device: Sham PEMF Device — Inactive device placed in the same manner as the active device; does not deliver pulsed electromagnetic fields
  Arms: Sham PEMF Device
Device: Ivivi Torino II PEMF Device — The PEMF device to be employed in this study is FDA cleared for "adjunctive use in the palliative treatment of postoperative pain and edema in superficial soft tissue" (510(k) number: K903675). The PEMF device will be taped over the affected breast and abdomen. The PEMF signal will consist of a 2 msec burst of 27.12 MHz sinusoidal waves repeating at 2 bursts/sec. The device will automatically provide a 15 minute treatment every 2 hours. Supplied by Ivivi Health Sciences, LLC.
  Other Names: Ivivi Torino II
  Arms: PEMF Device

SUMMARY:
Pedicled transverse rectus abdominus myocutaneous (TRAM) flaps are the most common post-mastectomy breast reconstructive surgeries that utilize the patient's tissue. The pedicled TRAM flap involves harvesting skin, fat, and muscle from the abdomen to create a new breast. TRAM flap complications include fat necrosis of the reconstructed breast, delayed wound healing, and abdominal bulge or hernia. Pain at the abdominal donor site is a major contributor to the need for four to five days of post-operative hospital stay. Pulsed electromagnetic field (PEMF) technologies have been useful as adjunctive therapy for the treatment of delayed union fractures, chronic wounds and post-operative pain. PEMF devices are economical and disposable, and can be incorporated unobtrusively in standard post-operative dressings. The investigators have recently reported, in a double-blind, placebo-controlled study on breast reduction, that post-op PEMF therapy produced a significant decrease in pain and pain medication use, along with a concomitant decrease in IL1-beta in the wound bed.

The proposed study seeks to determine whether similar results will be obtained after a significantly more extensive surgical procedure, like the TRAM flap. Patients scheduled for pedicled TRAM flap breast reconstruction of a single breast immediately following mastectomy will be enrolled in this double-blind, placebo-controlled, randomized study. Subjects will be assigned to one of two groups: a treatment group with active PEMF devices and a placebo group with sham devices that deliver no PEMF. PEMF and sham devices will be taped over both the breast reconstruction and abdominal donor sites. Patients will keep the devices in place for their hospital stay and for a total of two weeks. The investigators hypothesize that subjects in the PEMF treatment group compared to placebo will have a faster reduction in pain, take less pain and nausea medications, have lower levels of IL1-beta in wound exudate, have a shorter hospital stay, and have less wound-healing complications.

DETAILED DESCRIPTION:
Operations will be performed by one of two plastic surgeons who perform this surgery in a similar manner. The entire unilateral rectus abdominis muscle will be harvested with fascial-sparing as part of the pedicled TRAM flap. The flap will be shaped and sutured to the chest site, and the abdominal fascial defect will be closed primarily, followed by a polypropylene mesh overlay. Two 10 mm Jackson-Pratt (JP) drains will be placed in the flap wound, and two JPs will be placed in the abdominal wound. Immediately after transfer of the extubated patient to the recovery room bed, study devices will be placed on the reconstructed breast and abdominal donor sites, and activated. In the treatment arm, the PEMF signal is automatically delivered every two hours for fifteen minutes while the patient is in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients who decide to have immediate unilateral TRAM flap breast reconstruction and are deemed candidates for this surgery. Patients who have undergone or will be undergoing sentinel lymph node or axillary lymph node dissection will be included.

Exclusion Criteria:

* Patients who are not candidates for TRAM flap reconstruction will be excluded. Specific reasons for a patient not to be a candidate will be determined by the surgeon, but may include patients who have minimal abdominal tissue, patients with multiple medical co-morbidities, patients who have had prior abdominal surgeries that preclude a pedicled operation, or patients who are morbidly obese.
* Additionally, patients who opt for a free TRAM flap or DIEP flap will be excluded since their abdominal donor site morbidity is different than a pedicled TRAM flap.
* Patients undergoing bilateral reconstruction will also be excluded, because of the more extensive nature of the surgery and donor-site morbidity, which might confound results.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rohde, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rohde C, Chiang A, Adipoju O, Casper D, Pilla AA. Effects of pulsed electromagnetic fields on interleukin-1 beta and postoperative pain: a double-blind, placebo-controlled, pilot study in breast reduction patients. Plast Reconstr Surg. 2010 Jun;125(6):1620-1629. doi: 10.1097/PRS.0b013e3181c9f6d3. PMID 20527063
- [Derived] Rohde CH, Taylor EM, Alonso A, Ascherman JA, Hardy KL, Pilla AA. Pulsed Electromagnetic Fields Reduce Postoperative Interleukin-1beta, Pain, and Inflammation: A Double-Blind, Placebo-Controlled Study in TRAM Flap Breast Reconstruction Patients. Plast Reconstr Surg. 2015 May;135(5):808e-817e. doi: 10.1097/PRS.0000000000001152. PMID 25919263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from medical offices of two participating plastic surgeons.
Groups:
- PEMF Device: Ivivi Torino II PEMF Device: The PEMF device to be employed in this study is FDA cleared for "adjunctive use in the palliative treatment of postoperative pain and edema in superficial soft tissue" (510(k) number: K903675). The PEMF device will be taped over the affected breast and abdomen. The PEMF signal will consist of a 2 msec burst of 27.12 MHz sinusoidal waves repeating at 2 bursts/sec. The device will automatically provide a 15 minute treatment every 2 hours.
Period: Overall Study
Arm/Group | Sham PEMF Device | PEMF Device
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham PEMF Device | PEMF Device | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (9.1) | 51.1 (9.7) | 52.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 25.1 (3.1) | 24.5 (3.4) | 24.8 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Measured by Visual Analog Scale
Description: We will record postoperative pain, as reported by the patient and quantified by a standardized visual analog scale (VAS), with written descriptions at 12 hours post-op and assess that pain level in comparison with previous timepoint pain levels, such as 1 hour post-op. The VAS pain scale ranges from 0 (no pain) to 10 (worst possible pain). Higher scores indicate more pain and lower scores indicate less pain. The mean VAS score at 12 hours is reported for each group, active or placebo.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham PEMF Device | PEMF Device
Number analyzed (Participants) | 16 | 16
units on a scale | 3.48 (0.61) | 1.67 (0.43)
Statistical Analysis 1: Comparison: Sham PEMF Device vs PEMF Device; Before the start of this study, a sample size analysis, assuming a clinically meaningful 50± 40 percent (mean ± SD) decrease in pain scores from pulsed electromagnetic field treatment, suggested that a minimum of 11 patients per group were needed; Test type: Superiority — Applies to primary and secondary outcomes: Data were analyzed using one-way analysis of variance, one-way repeated measures analysis of variance, t test, or Mann-Whitney rank sum test, as appropriate. (SigmaStat 3.5; Systat Software, Inc., San Jose, Calif.). Intention-to-treat using last value carried forward was used for missing data; p < 0.01, ANOVA

2. Secondary Outcome: Number of Narcotic Pain Medications
Description: We will record the amount of pain medication used at twelve hour intervals for the duration of the hospital stay. Pain medications will be converted to oxycodone/acetaminophen equivalents for statistical analysis
Time Frame: 24 hours
Population: data reported at 24 hours postop
Measure: Mean (Standard Deviation); unit: pills
Arm/Group | Sham PEMF Device | PEMF Device
Number analyzed (Participants) | 16 | 16
pills | 34 (2.8) | 20 (1.8)

3. Secondary Outcome: Levels of Cytokines
Description: Concentration of the cytokines IL1-beta in the wound bed. Exudates will be collected from standard Jackson-Pratt #10 drains until the patient is discharged. IL1-beta is an early central proinflammatory cytokine that induces cyclooxygenase, an enzyme responsible for prostaglandin synthesis. A decrease in IL1-beta correlates with a decrease in pain. Cytokines and growth factors may contribute to more rapid post-op pain reduction and healing.
Time Frame: 24 hours
Population: data reported at 24 hours postop
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Sham PEMF Device | PEMF Device
Number analyzed (Participants) | 16 | 16
pg/ml | 320 (36) | 168 (17)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the time period in which the PEMF device was in place post-operatively, usually less than 7 days post-op.
Arm/Group | Sham PEMF Device | PEMF Device
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No